CLINICAL TRIAL: NCT01083589
Title: Phase II Study of Imatinib Mesylate and Docetaxel in Pretreated Patients With Metastatic NSCLC
Brief Title: Imatinib Mesylate and Docetaxel in Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0726
Record Dates: First submitted 2010-03-08; First posted 2010-03-10 (Estimated); Last update posted 2012-01-11 (Estimated); Status verified 2012-01

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Lung Cancer; Metastatic NSCLC; Tumor; Imatinib Mesylate; Gleevec; Docetaxel; Taxotere
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Neoplasms | interventions — Imatinib Mesylate; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Imatinib Mesylate + Docetaxel (Experimental): Imatinib Mesylate (Gleevec) Oral 400 mg daily + Docetaxel (Taxotere) 60 mg/m2 over 1 hour intravenous infusion repeated every 21 days.
  Interventions: Drug: Imatinib Mesylate; Drug: Docetaxel

INTERVENTIONS:
Drug: Imatinib Mesylate — Oral 400 mg daily
  Other Names: Imatinib; Gleevec; STI571; NSC-716051
Drug: Docetaxel — 60 mg/m2 over 1 hour intravenous infusion repeated every 21 days.
  Other Names: Taxotere

SUMMARY:
The goal of this clinical research study is to learn how effective the combination of the drugs imatinib mesylate (Gleevec®) and docetaxel (Taxotere®) is in treating non-small cell lung cancer (NSCLC). The safety and tolerability of this drug combination will also be studied.

DETAILED DESCRIPTION:
Imatinib mesylate is a medication that blocks certain proteins important in the development of cancer. Docetaxel is a drug that is designed to target and destroy cancer cells.

If you are found to be eligible to take part in this study, you will take 4 imatinib mesylate tablets by mouth once a day. Docetaxel will be given through a vein in your arm on the first day of each treatment cycle for a total of 6 cycles. The infusion will take 1 hour. A treatment cycle on this study is 21 days.

You will need to take steroids (dexamethasone) before receiving docetaxel to try to prevent fluid accumulation and hypersensitivity reactions. The dexamethasone will come in a pill form to be taken every 12 hours for 3 days starting the day before chemotherapy. You will also receive additional dexamethasone by vein before the docetaxel is given.

After you complete 6 treatment cycles, you will continue to take 4 imatinib mesylate tablets each day until your cancer gets worse, or you experience unacceptable side effects, or you withdraw from the study.

While on this study, you will have a physical exam every 3 weeks. During the first 5 weeks of the study, you will have blood tests each week. About 3 teaspoons of blood will be drawn each time. After the first 5 weeks, you will have blood tests (3 teaspoons each) at the beginning of each treatment cycle. In addition, your tumor will be measured by a CT or MRI scan every 6 weeks.

You must agree not to use herbal remedies or other over-the-counter therapies (e.g., shark cartilage) during treatment.

If you develop any unacceptable symptoms or changes in your laboratory tests, your treatment may be delayed and/or the dose decreased until the symptoms are gone. It may even be necessary to stop your treatment. Your doctor will inform you of any changes in your dosing schedule or in the doses of your medication after he/she evaluates you in the clinic.

After treatment ends, you will have a follow-up visit at the clinic. At this visit, you will have a complete physical exam, including blood (about 3 teaspoons) and urine tests. You will also have a CT scan to measure the size of the tumor in your body.

This is an investigational study. Imatinib mesylate is FDA approved for the treatment of leukemia. Docetaxel is FDA approved for the treatment of breast, prostate, and NSCLC. Up to 50 patients will take part in this study. All will be enrolled at UTMDACC.

ELIGIBILITY:
Inclusion Criteria:

1. An written, voluntary informed consent form must be completed prior to beginning any study procedure.
2. Patients >/= 18 years of age.
3. Histologically documented diagnosis of non-small cell lung cancer.
4. At least one measurable site of disease that is amenable to biopsy. Lesion must be at least 20 mm in the longest diameter by spiral computed tomography (CT) or 20 mm with conventional techniques according to RECIST. Lesion must not have been previously irradiated.
5. Performance status 0-1 (Eastern Cooperative Oncology Group (ECOG))
6. Patients must have adequate hepatic, renal, and bone marrow function, defined as the following: (1) total bilirubin < 1.5 * upper limit of normal (ULN); (2) serum glutamic oxaloacetic transaminase (SGOT) and serum glutamic pyruvic transaminase (SGPT) < 2.5 * UNL; (3) creatinine < 1.5 * ULN; (4) ANC > 1.5 * 10^9/L; (5) platelets > 100 * 10^9/L.
7. Female patients of childbearing potential must have negative pregnancy test within 7 days before initiation of study drug dosing. Postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential. Male and female patients of reproductive potential must agree to employ an effective barrier method of birth control throughout the study and for up to 3 months following discontinuation of study drug.
8. Patients who have received one prior systemic chemotherapy treatment (not including biologic agents e.g. gefitinib, lonafarnib).
9. Patients who were originally diagnosed with earlier stage Non-small-cell lung carcinoma (NSCLC) & were treated with curative intent (i.e. pts who have received induction chemotherapy (platinum-based doublet) prior to definitive radiation or surgery) but then develop recurrent or metastatic disease & are then treated with a platinum-based doublet for frontline metastatic therapy are still eligible for this study. This is as long as they have not been exposed to docetaxel during any point of their therapy. Once patients have been diagnosed with metastatic or recurrent disease, they may only have received one platinum-based therapy.

Exclusion Criteria:

1. Patient has received any other investigational agents within 30 days of first day of study drug dosing.
2. Patient is < 5 years free of another primary malignancy except: if the other primary malignancy is not currently clinically significant nor requiring active intervention, or if other primary malignancy is a basal cell skin cancer or a cervical carcinoma in situ. Existence of any other malignant disease is not allowed.
3. Patient with Grade III/IV cardiac problems as defined by the New York Heart Association Criteria. (i.e., congestive heart failure, myocardial infarction within 6 months of study)
4. Female patients who are pregnant or breast-feeding.
5. Patient has a severe and/or uncontrolled medical disease (i.e., uncontrolled diabetes, chronic renal disease, or active uncontrolled infection).
6. Patient has a known untreated or unstable brain metastasis.
7. Patient has known chronic liver disease (i.e., chronic active hepatitis, and cirrhosis).
8. Patient has a known diagnosis of human immunodeficiency virus (HIV) infection. HIV patients are at much greater risk of infection when receiving highly myelosuppressive agents (docetaxel and imatinib) and for safety reasons are not eligible for this trial.
9. Patient received chemotherapy within 4 weeks (6 weeks for nitrosourea or mitomycin-C) prior to study entry, unless the disease is rapidly progressing.
10. Patient previously received radiotherapy to >/= 25 % of the bone marrow
11. Patient had a major surgery within 2 weeks prior to study entry.
12. Patient with any significant history of non-compliance to medical regimens or with inability to grant reliable informed consent.
13. Patients must agree not to use herbal remedies or other over-the-counter biologics (i.e. shark cartilage)
14. History of hypersensitivity to docetaxel or other taxane therapy.
15. History of severe hypersensitivity reaction to drugs formulated with polysorbate 80.
16. Prior exposure to imatinib mesylate.
17. Prior exposure to docetaxel systemic therapy for this NSCLC malignancy.
18. Patient treated with more than 1 prior systemic chemotherapy (not including biologic agents e.g. gefitinib, lonafarnib)
19. Participation in an investigational trial within the past 30 days.
20. Patients taking therapeutic levels of warfarin. However, patients receiving 1 mg daily for catheter related anticoagulation are eligible for the study.
21. Prior pericardial effusion requiring intervention such as pericardiocentesis or pericardial window.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2005-01; Primary Completion 2007-10 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Patient Response Rate | Baseline and with each 3 week cycle
  Response rate to new regimen defined as the percentage of complete or partial response within the total number of patients treated. Treatment response assessed by Response Evaluation Criteria In Solid Tumors (RECIST) criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Anne S. Tsao, MD, Study Chair — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org